CLINICAL TRIAL: NCT01790256
Title: A Multi-center Prospective, Blinded, Randomized Crossover Study to Compare the Cerêve Sleep System at Two Different Temperatures in Primary Insomnia Patients
Brief Title: Comparison of Two Temperatures to Treat Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cereve, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Cereve CIP-003
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cereve Sleep System at 14-16 degrees C. (Active Comparator): Active
  Interventions: Device: Cereve Sleep System at 14-16 degrees C
- Cereve Sleep System at 30 degrees C (Active Comparator): Active
  Interventions: Device: Cereve Sleep System at 30 degrees C

INTERVENTIONS:
Device: Cereve Sleep System at 30 degrees C
  Arms: Cereve Sleep System at 30 degrees C
Device: Cereve Sleep System at 14-16 degrees C
  Arms: Cereve Sleep System at 14-16 degrees C.

SUMMARY:
Insomnia patients demonstrate subjective and physiological hyperarousal. The Cereve Sleep System has been proposed as a clinical treatment to reverse this hyperarousal in insomnia patients. The current study is a two dose study to determine the optimal temperature for the Cereve Sleep System. Primary outcome measures include EEG sleep measured sleep latency and sleep efficiency.

ELIGIBILITY:
Inclusion Criteria:

Age >/= 22

Diagnosis of insomnia that meets criteria for DSM IV diagnosis of primary insomnia and International Classification of Sleep Disorders (ICSD)general insomnia criteria and RDC insomnia disorder criteria

Subjects must remain alcohol-free and avoid drugs that could affect sleep during the study.

>14 on the Insomnia Severity Index

Sleep -Wake diaries demonstrate sleep efficiency <85% on at least 50% of nights

Exclusion Criteria:

Neuropsychiatric disorders that may independently affect sleep, brain function or cognition, such as current major syndromal psychiatric disorders, including DSM-IV mood, anxiety, psychotic, and substance use disorders.

Specific exclusionary diagnoses include major depressive disorder, dysthymic disorder, bipolar disorder, panic disorder, obsessive compulsive disorder, generalized anxiety disorder, any psychotic disorder, and any current substance use disorder.

Unstable medical conditions Raynaud's Disease

Irregular sleep schedules including shift workers;

A latency to persistent sleep < 15 on either the sleep disorder screening night or the baseline PSG sleep night;

A sleep efficiency > 85% on either the sleep disorder screening night or the baseline PSG sleep night;

An AHI (apnea hypopnea index) > 10 and/or a periodic limb movement arousal index (PLMAI) > 15 from SN1

Body Mass Index >34

Use of medications known to affect sleep or wake function

Consumption of more than one alcoholic drink per day, or more than 7 drinks per week prior to study entry.

Caffeinated beverages > 4/day or the equivalent of more than 4 cups of coffee Unable to read or understand English

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Polysomnographically determined sleep latency as changed from baseline measures | 1-2 weeks
  Polysomnographically determined sleep parameters
Poloysomnographically determined sleep efficiency as changed from baseline measures | 1-2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lankford, PhD, Principal Investigator — Sleep Center of Georgia; Russell Rosenberg, PhD, Principal Investigator — Neurotrials; Leon Rosenthal, MD, Principal Investigator — Sleep Medicine Associates of Texas; David Mayleben, PhD, Principal Investigator — Community Research; Paul Wylie, MD, Principal Investigator — Preferred Research Partners; Mark Muehlbach, PhD, Principal Investigator — Clayton Sleep Institute; David Seiden, MD, Principal Investigator — Broward Research Group; Timothy Grant, MD, Principal Investigator — Miami Research Associates; Neil Feldman, MD, Principal Investigator — Clinical Research Group of St. Petersburg
Locations (9):
- United States (9):
  - Paul Wylie, Little Rock, Arkansas
  - Timothy Grant, Miami, Florida
  - David Seiden, Pembroke Pines, Florida
  - Neil Feldman, St. Petersburg, Florida
  - Alan Lankford, Atlanta, Georgia
  - Russell Rosenberg, Atlanta, Georgia
  - David Mayleben, Crestview Hills, Kentucky
  - Mark Muehlbach, St Louis, Missouri
  - Leon Rosenthal, Dallas, Texas